CLINICAL TRIAL: NCT03772548
Title: Functional, Structural, and Metabolic Central Nervous System Changes Following Damage of the Central Nervous System
Brief Title: CNS Changes Following SCI
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-00937 - SCI
Record Dates: First submitted 2018-11-21; First posted 2018-12-11 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with spinal cord injury
  Interventions: Diagnostic Test: MRI
- Healthy subjects
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — We will examine acute (<4 weeks post SCI) to chronic (>6 months post SCI) patients using functional, structural, and metabolic MRI in both the brain and the spinal cord.
  Groups: Patients with spinal cord injury
Diagnostic Test: MRI — We will examine healthy control participants using functional, structural, and metabolic MRI in both the brain and the spinal cord.
  Groups: Healthy subjects

SUMMARY:
The objective of this study is to better understand the structural and functional changes that the central nervous system (CNS) undergoes following spinal cord injury and how these changes relate to clinical measures. Both macroscopic and microscopic changes of the brain and the spinal cord will be examined in SCI patients and compared to healthy controls. In terms of structural plasticity, we aim to identify MR biomarkers that allow predicting the course of the patient's neurological status and accurately describe the course of the disease and the recovery. Importantly, we aim to investigate which factors scale the patients' symptoms. In terms of functional plasticity, we will combine fMRI with behavioural testing to understand which clinical and behavioural determinants drive functional hand representations in the primary somatosensory and motor cortices to be maintained and which determinants drive reorganisation of functional representations following sensory input loss. We will further investigate the contribution of brainstem reorganisation to plasticity observed at the cortical level and, by doing so, aim to better understand the mechanistic underpinnings of functional reorganisation.

ELIGIBILITY:
Inclusion Criteria - Patients:

* Age 18-75
* Traumatic or non-traumatic spinal cord injury (para- and tetraplegia)
* Acute (<4 weeks post SCI) to chronic SCI (> 6 months post SCI)
* Signed informed consent

Exclusion Criteria - Patients:

* Contraindications to magnetic resonance imaging
* Neurological impairment of body function impairments not induced by spinal cord injury
* BMI > 40
* Pregnancy
* Claustrophobia

Inclusion Criteria - Healthy subjects:

* Age 18-75
* Signed Informed consent

Exclusion Criteria - Healthy subjects:

* Contraindications to magnetic resonance imaging
* Pregnancy
* Neurological illness
* Impairment of body function induced by a spinal cord injury
* Claustrophobia
* BMI > 40

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with spinal cord injury and healthy subjects.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2018-07-18 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Conventional magnetic resonance imaging (MRI) parameter | Up to 50 weeks
  Structural characteristics in the brain and cervical spinal cord are assessed in acute to chronic spinal cord injury (SCI) patients using conventional MRI and compared to healthy controls

SECONDARY OUTCOMES:
Magnetic resonance spectroscopy (MRS) parameter | Up to 50 weeks
  Metabolic parameters are assessed in acute to chronic SCI patients using MRS in the brain and cervical spinal cord and compared to healthy controls
Change of functional MRI (fMRI) parameter between 2 to 4 time points | Up to 50 weeks
  Change of brain activities is assessed between 2 to 4 time points using fMRI during resting-state or a specific task in acute to chronic SCI patients and compared to healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Freund, Prof. Dr., Principal Investigator — University of Zurich
Locations (1):
- Universitätsklinik Balgrist, Zurich, Switzerland

REFERENCES:
- [Derived] Kikkert S, Pfyffer D, Verling M, Freund P, Wenderoth N. Finger somatotopy is preserved after tetraplegia but deteriorates over time. Elife. 2021 Oct 19;10:e67713. doi: 10.7554/eLife.67713. PMID 34665133